CLINICAL TRIAL: NCT03681470
Title: An Open-label Study to Investigate the Efficacy and Tolerability of Aczone Gel, 7.5% in the Treatment of Acne Vulgaris in Men and Women With Skin of Color
Brief Title: Aczone Gel 7.5% in the Treatment of Acne Vulgaris in Patients With Skin of Color
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Saakshi Khattri, Assistant Professor, Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2662; HSM# 17-01277 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Acne Vulgaris
Keywords: skin of color; acne; skin diseases
MeSH Terms: conditions — Acne Vulgaris; Skin Diseases | interventions — Dapsone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Acne Vulgaris (Experimental): Acne Vulgaris in Patients With Skin of Color
  Interventions: Drug: Aczone Gel

INTERVENTIONS:
Drug: Aczone Gel — Aczone Gel 7.5%
  Other Names: Dapsone

SUMMARY:
Acne vulgaris is a common skin disease characterized by inflammatory papules, pustules, and comedones that is prevalent in men and women of color. Research has demonstrated that Aczone ® (dapsone) gel, 7.5% used once daily is effective, safe, and well-tolerated for the treatment of acne in both men and women; however, limited data is available regarding its efficacy and safety in skin of color (SOC). The current study aims to investigate the therapeutic impact of Aczone gel 7.5% in SOC males and females ages 18 and older with acne vulgaris. The study will also evaluate the impact of Aczone ® gel on hyperpigmentation and PIH of the face.

DETAILED DESCRIPTION:
Acne vulgaris is a common skin disease characterized by inflammatory papules, pustules, and comedones that is prevalent in men and women of color. In fact, acne is the most common dermatologic diagnosis made in SOC populations. Although individuals of all skin types can develop acne vulgaris, there are important differences in darker skin types that are important to consider when choosing an optimal treatment.

Complications from acne are of great concern in this population, as keloids, hypertrophic scars, and post-inflammatory hyperpigmentation (PIH) are more common in skin of color. PIH may last for weeks to months and, in many cases, is more troublesome to patients than the acne itself. Overall, facial acne and its sequelae have a greater impact on perception of appearance, negative emotions, and social functioning in women of color than white women.

Dapsone is a sulfone compound with anti-inflammatory properties that has been shown to be effective in the treatment of acne vulgaris in SOC. Aczone ® (dapsone) gel, 5% administered twice daily has been associated with significant improvement in overall acne severity, acne signs, and impact on quality of life in women of color. Two phase III trials of a newer formulation of Aczone ® (dapsone) gel, 7.5% used once daily demonstrated that this product is effective, safe, and well-tolerated for the treatment of acne in both men and women; however, limited data is available regarding its efficacy and safety in SOC.

Further, some investigators of the phase IV study on the safety and efficacy of dapsone gel 5% in SOC anecdotally reported improvement in hyperpigmentation over 12 weeks, although this was not a planned efficacy outcome. Further research is needed on the potential effects of dapsone gel on hyperpigmentation and PIH in SOC.

The current study will investigate the therapeutic impact of Aczone gel 7.5% in SOC males and females ages 18 and older with acne vulgaris. The study will also evaluate the impact of Aczone gel on post-inflammatory hyperpigmentation using the Postacne Hyperpigmentation Index (PAHPI) and mexameter-measured melanin index (MI).

ELIGIBILITY:
Inclusion Criteria:

* Provide written, signed and dated informed consent prior to initiating any study-related activities.
* Male or female subjects who are ≥ 18 years of age
* Subjects with Fitzpatrick Skin Type IV, V, or VI
* Subjects with moderate to severe acne as defined by investigator- assessed Global Acne Assessment Score (GAAS) of 3 or 4 at screening
* Facial acne vulgaris with 20 to 50 (inclusive) inflammatory lesions and 30 to 100 (inclusive)non inflammatory lesion
* Stable non-progressive or regressive acne vulgaris in the investigator's opinion
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. A female is considered not to be of childbearing potential if she is post-menopausal with at least 12 consecutive months of amenorrhea or has undergone surgical sterilization. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

* Must be in general good as judged by the Investigator
* Subject is willing to avoid excessive or prolonged exposure of the treated skin to ultraviolet light (i.e. sunlight, tanning beds) throughout the study
* Subject is willing to follow study instructions and complete study assessments without assistance and is likely to complete all required visits

Exclusion Criteria:

* Diagnosis of other dermatologic diagnosis that, in the opinion of the investigator, would interfere with diagnosis, examination, or treatment of the studied condition (i.e. psoriasis, atopic dermatitis, lupus, dermatomyositis, seborrheic dermatitis, perioral dermatitis, etc.)
* Subjects with severe cystic acne, acne conglobate, acne fulminans, or secondary acne (chloracne or drug-induced acne)
* Uncontrolled systemic disease(s) that, in the opinion of the investigator, would put the patient at significant risk if enrolled in the study or would interfere with subject's participation in the study
* Subjects with a history of clinically significant hemolysis, anemia, or enteritis (regional enteritis, ulcerative colitis, pseudomembranous colitis, antibiotic-associated colitis)
* Subjects with allergy or sensitivity to the study drug or its components
* Subjects who have not complied with the proper wash-out periods:

  * Topical anti-inflammatory medications, salicylic acid, corticosteroids, antibiotics, antibacterials, peroxide-containing products, or retinoids within 2 weeks of baseline
  * Systemic antibiotics, corticosteroids, antimalarials or oral dapsone within 4 weeks of baseline Other anti-acne medication, including isotretinoin or spironolactone, within 6 months of baseline
  * Chemical peels or other facial acne procedures (laser therapy, light therapy) within 3 months of baseline
  * Treatment with botulinum toxin of any serotype in the face within 6 months of baseline
  * Estrogens/Birth control pills must have been started ≥ 90 days prior to baseline and use must be continued during the study without alteration or discontinuation.
  * Pregnant or breast feeding.
  * Subjects with evidence of alcohol or substance abuse.
  * Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saakshi Khattri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
IDP will be shared with Allergan
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available upon completion of the study and will remain available until final publication of the data
Access Criteria: Will only be shared with staff of Allergen directly involved with oversight of clinical study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Acne Vulgaris
Started | 20
Completed | 12
Not Completed | 8
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 0
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 12 in Global Acne Assessment Score (GAAS)
Description: GAAS assesses acne severity on a 5-point score:
  0 - None: No evidence of facial acne vulgaris.
  1. - Minimal: Few noninflammatory lesions are present; a few inflammatory lesions (papules/pustules) may be present; no nodulo-cystic lesions present.
  2. - Mild: Several to many noninflammatory lesions are present; a few inflammatory lesions are present; no nodulo-cystic lesions present.
  3. - Moderate: Many noninflammatory and inflammatory lesions are present; no nodulo-cystic lesions are present.
  4. - Severe: Significant degree of inflammatory disease; papules and pustules are a predominant feature; a few nodulo-cystic lesions are present (no more than 2)
Time Frame: baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
score on a scale | -0.86 (0.66)

2. Secondary Outcome: Change From Baseline in Global Acne Assessment Score (GAAS) at Week 4, 18 and 24
Description: Change from baseline at week 4, week 18 and week 24.
  GAAS assesses acne severity on a 5-point score:
  0 - None: No evidence of facial acne vulgaris.
  1. - Minimal: Few noninflammatory lesions are present; a few inflammatory lesions (papules/pustules) may be present; no nodulo-cystic lesions present.
  2. - Mild: Several to many noninflammatory lesions are present; a few inflammatory lesions are present; no nodulo-cystic lesions present.
  3. - Moderate: Many noninflammatory and inflammatory lesions are present; no nodulo-cystic lesions are present.
  4. - Severe: Significant degree of inflammatory disease; papules and pustules are a predominant feature; a few nodulo-cystic lesions are present (no more than 2)
Time Frame: baseline and week 4, week 18, and week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
score on a scale
  Baseline and Week 4 | -0.35 (0.49)
  Baseline and Week 18 | -1.0 (0.77)
  Baseline and Week 24 | -1.2 (0.79)

3. Secondary Outcome: Change From Baseline in Post Acne Hyperpigmentation Index (PAHPI) at Weeks 12, 18 and 24
Description: Change from baseline at weeks 12, 18, and 24.
  PAHPI will be scored using the following formula:
  Weighted Total PAHPI = S (lesion size) + I (lesion intensity) + N (lesion number). Total PAHPI Score can range from 6-22, with higher number indicating more pigmentation.
Time Frame: baseline and week 12, 18, and 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
score on a scale
  baseline and week 12 | -1.7 (1.77)
  baseline and week 18 | -2.22 (2.28)
  baseline and week 24 | -3 (2.58)

4. Secondary Outcome: Change From Baseline in Melanin Index (MI) of Target Lesion at Weeks 12, 18 and 24
Description: A narrowband reflectance spectrophotometer (mexameter MX-16) will be used to measure the degree of pigmentation of involved and adjacent uninvolved skin of one representation facial PIH lesion.
  The mexameter contains 16 light emitting diodes arranged circularly that emit light at wavelengths of 568nm (green), 660nm (red), and 880nm (near infrared). The machine then measures the amount of light absorbed and reflected by the skin to measure the melanin content (melanin index or "M" - red and near infrared light).
  There is no minimum or maximum to this index. Higher melanin index indicates more melanin content in the skin. Higher or increase MI indicates poorer health outcomes.
Time Frame: baseline and week 12, 18 and 24
Measure: Mean (Standard Deviation); unit: Melanin Index (M)
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
Melanin Index (M)
  baseline and week12 | 0.22 (13.94)
  baseline and week 18 | -2.33 (8.94)
  baseline and week 24 | -48.5 (77.22)

5. Secondary Outcome: Number of Subjects With Score of 0 or 1 on ASIS "Dark Spot" Score at Weeks 4, 12, 18 and 24
Description: The participant assesses signs of acne vulgaris using the Acne Symptom and Impact Scale (ASIS). The sign domain is a composite of 9 items of the 17 items on the overall scale. Each of the items is answered on a 5-point scale: 0 (best) to 4 (worst). Total possible score of 0 to 68. Higher scores indicate the presence of more severe symptoms and poorer outcomes on acne health-related quality of life.
Time Frame: week 4, 12, 18, and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
Participants
  week 4 | 2
  week 12 | 2
  week 18 | 4
  week 24 | 7

6. Secondary Outcome: Number of Subjects With GAAS of 0 (None) or 1 (Minimal) at Weeks 4, 12, 18, 24
Description: The change in the proportion of subjects with GAAS scores equal to 0 (or 1) from baseline.
  GAAS assesses acne severity:
  0 - None: No evidence of facial acne vulgaris.
  1 - Minimal: Few noninflammatory lesions are present; a few inflammatory lesions (papules/pustules) may be present; no nodulo-cystic lesions present.
Time Frame: Week 4, 12, 18 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
Participants
  Week 4 | 0
  Week12 | 2
  Week 18 | 3
  Week 24 | 4

7. Secondary Outcome: Percent Change From Baseline in All Lesion Counts (Inflammatory, Noninflammatory, and Total) at Weeks 4, 12, 18, and 24
Time Frame: Baseline, Week 4, 12, 18, and 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Patients With Acne Vulgaris
Number analyzed (Participants) | 12
percent change
  Baseline and week 4 | -29 (19)
  Baseline and week 12 | -46 (24)
  Baseline and week 18 | -55 (23)
  Baseline and week 24 | -53 (31)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Patients With Acne Vulgaris
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Acne Vulgaris (N=20)
Dry patches of skin (Skin and subcutaneous tissue disorders) | 1
Traction alopecia (Skin and subcutaneous tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Upper respiratory infection (Infections and infestations) | 2
Syncope (Nervous system disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Vocal cord fatigue (General disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Common cold (Infections and infestations) | 1
Post inflammatory hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Worsening post inflammatory hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Rough facial skin (Skin and subcutaneous tissue disorders) | 1
Right hand burn (General disorders) | 1
COVID-19 (Infections and infestations) | 1
left hand burn (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03681470/Prot_SAP_000.pdf